CLINICAL TRIAL: NCT05404932
Title: Management of Recurrent and Progressive Ligneous Conjunctivitis Due to Plasminogen Deficiency. An N of One Clinical Trial of Topical Administration of Allogenic Plasma to Affected Eye
Brief Title: Treatment of Ligneous Conjunctivitis in Children With Plasminogen Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Blood Services (Other)
Responsible Party: Principal Investigator, Sarah Tehseen, Principle Investigator, Assistant Professor of Pediatric Hematology and transfusion medicine, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USASK0511ST
Record Dates: First submitted 2022-05-12; First posted 2022-06-03 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Plasminogen Deficiency
MeSH Terms: conditions — Congenital Plasminogen Deficiency

STUDY DESIGN:
Intervention Model Description: Only one patient (and their family) with laboratory diagnosis of plasminogen deficiency and ligneous conjunctivitis will be enrolled in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (aliquoted plasma application into the conjunctiva) (Experimental): This is the only arm of the study. The intervention is administration of aliquoted plasma provided by Canadian Blood Services in eye droppers (3 ml aliquots in 7 ml vials) in the patient's conjunctiva.
  The duration of therapy can be 2 to 6 months depending on response The intra-ocular drops will be administered every 1-5 hours daily in the affected eye based on disease severity and may be repeated
  Interventions: Drug: Aliquoted allogeneic donor plasma in patient's conjunctiva

INTERVENTIONS:
Drug: Aliquoted allogeneic donor plasma in patient's conjunctiva — 1-2 drops of allogenic aliquoted plasma to affected eye every 1-5 hours per day based on disease severity to be weaned down based on clinical response Administration period: Two to Six months. This may be repeated based on recurrence/worsening of conjunctivitis

SUMMARY:
Congenital plasminogen deficiency causes impaired wound healing and growth of pseudomembranous lesions over multiple parts of the body. The most common lesions involve eyes and are known as Ligneous conjunctivitis. These can cause scarring of the sclera, vision loss and even blindness. These pseudomembranous lesions are recur after surgical excisions, administration of intra-ocular cyclosporine, autologous serum drops or corticosteroids.

Clinical data shows that these growths do not worsen and do not recur after administration of plasminogen (either as concentrate or as plasma) in the eyes, locally or intravenously.

As plasminogen is not available as concentrate, we are using aliquoted allogenic plasma provided by Canadian Blood Services for intra-ocular application. These will be applied to eyes multiple times a day for a period of 2 to 6 months depending on disease severity and patient response. These may be used again if ligneous conjunctivitis recurs.

The patient will be followed for a period of 2 years at least. All serious adverse events will be reported to Canadian Blood Services and Health Canada as appropriate.

DETAILED DESCRIPTION:
This study will enroll one patient with recurrent ligneous conjunctivitis at University of Saskatchewan, Saskatchewan Health Authority in Saskatoon.

BACKGROUND:

Congenital plasminogen deficiency is an extremely rare autosomal recessive disorder that leads to formation of extravascular fibrin rich pseudomembranes in various organ systems including central nervous system, gastrointestinal, respiratory and otopharyngeal tracts (1, 2, 3). Conjunctival involvement in the form of recurrent woody growths underneath the eyelid (ligneous conjunctivitis) is the most common manifestation (5, 6). The symptoms are most severe in infants and children, where it may lead to central nervous system (CNS) hydrocephalus, respiratory failure or blindness, depending on the organ system involved (3,4)

The conjunctival pseudomembranes recur after excision and show a poor response to topical steroids, cyclosporine, or autologous serum administration. These lesions can lead to conjunctival scarring, ptosis, loss of visual acuity and ultimately blindness5,6.

Plasminogen replacement (in the form of topical drops of plasminogen concentrate or allogenic plasma) has proven to be the most effective modality in preventing growth of these lesions and is required by most patients to prevent end organ damage.

RATIONALE:

More than 200 cases of plasminogen deficiency have been reported in literature.(14) Plasminogen replacement (in the form of intraocular drops of plasminogen concentrate or donor plasma) has proven to be the most effective modality in preventing growth of these lesions and is required by most patients to prevent end organ damage (7-20).

Plasminogen concentrate is not an option as plasminogen concentrates are not available in Canada. There is one company that produces plasminogen concentrate in North America that is currently not supplying any products on compassionate basis and there are no open clinical trials. Another company (Kedrion) produces it in Italy though it is also not providing on compassionate basis. It is significantly cost prohibitive. Cost: 2800 Euros per ml of concentrate. The product needs to be applied to affected conjunctiva 3-8 times per day for ~3-12 months.

Heparin Therapy alone: Case report data shows utilization of Heparin therapy alone for ligneous conjunctivitis in children which led to orbital inflammation and cellulitis with only partial control of lesion (2).

Sustained control of these lesions has only been achieved with administration of plasminogen (Intravenous [IV]/local) or plasma (as a source of plasminogen) alone or in conjunction with other therapies (such as membrane resection, heparin etc (7-13), (15-20).

TRIAL OBJECTIVES AND PURPOSE:

1. Determine safety of topical administration of aliquoted allogeneic plasma to the affected eye.
2. Determine efficacy of topical administration of aliquoted allogenic plasma.

TRIAL TREATMENTS:

The allogenic plasma will be aliquoted into 3 ml aliquots and placed in 7 ml vials/bottles. The vials will be frozen at -18 degree Celsius or lower temperature. To administer, the vial/bottle will be warmed to room temperature (15-30 degree Celsius). 1-2 drops of aliquoted donor plasma will be administered to the affected eye every 1-5 hours per day daily at maximum. The administration of plasma drops can change in frequency based on the clinical assessment of ligneous conjunctivitis and response to therapy.

STUDY DURATION

The treatment administration period will be 2 to 6 months. The duration of study participation, including follow-up, will be approximately 24 months.

STUDY VARIABLES

The following data will be collected for this study:

1. Size of pseudomembranous conjunctival lesion
2. Visual acuity of the affected eye
3. Development of strabismus or other visual defects in affected eye
4. Medical history
5. Physical exam
6. Blood group (ABO, RhD) and antibody screen results
7. Details of any adverse events

All data will be collected on the data collection form. The participant's medical record will be considered to be a source document for the medical history. The lab report will be considered the source document for the lab tests.

STOPPING RULES AND DISCONTINUATION CRITERIA

Criteria for discontinuation

1. Patient does not want to continue the study
2. Patient has a significant adverse reaction to plasma drops
3. Patient has no response to therapy after 6 months of intervention. This is defined as:

   1. No change in the size of pseudomembranes after 6 months of topical allogenic plasma administration performed according to recommendations (with/without surgical excision)
   2. Increase in the size of pseudomembranous lesions despite recommended use of aliquoted allogenic plasma
   3. Development of new pseudomembranous lesions in the eye receiving topical allogenic plasma
4. More effective therapies (liquid plasminogen concentrate IV/Intra-ocular) become available in Canada
5. Plasma drops can no longer be provided

MONITORING OF PARTICIPANT COMPLIANCE

Participant compliance will be assessed by maintaining adequate drug dispensing logs and return records. Participants will be asked to return all unused study drug in the provided container at each visit as a measure of drug accountability and patient compliance.

ASSESSMENT OF SAFETY

Safety Parameters include:

1. Direct clinical monitoring of patient during initial 5 intra-ocular plasma administrations
2. Communication with the patient and family at least on a weekly basis while receiving intra-ocular plasma.
3. Source plasma collected from donors who are negative for transfusion transmissible infections
4. Source plasma cultured before release to facility to ensure no bacterial contamination
5. Clear guidance to parents about situations where plasma administration should be stopped, and clinical care accessed.
6. Communication to the pediatric hematology service available 24/7 in case of any issues with plasma administration
7. Close liaison with pediatric ophthalmologist who will also monitor response and potential complications

ADVERSE EVENTS and MITIGATION STRATEGIES

According to the ICH guideline for Good Clinical Practice, an adverse event is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

Serious Adverse Events

A serious adverse event is any adverse event that meets any of the following criteria:

1. Fatal (i.e., the adverse event actually causes or leads to death) 2. Life threatening (i.e., the adverse event, in the view of the investigator, places the patient at immediate risk of death). This does not include any adverse event that had it occurred in a more severe form, or was allowed to continue, might have caused death 3. Requires or prolongs inpatient hospitalization 4. Results in persistent or significant disability/incapacity (i.e., the adverse event results in substantial disruption of the patient's ability to conduct normal life functions) 5. Congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug 6. Significant medical event in the investigator's judgment (e.g., may jeopardize the patient or may require medical/surgical intervention to prevent one of the outcomes listed above). RISK MITIGATION STRATEGIES

1. Loss of patient privacy and confidentiality:

   1. All patient information will be recorded in hospital electronic medical record systems which have adequate protections in place to prevent unauthorized spread of patient information.
   2. The data collected for clinical trial will be maintained in University Operated Redcap which will be password protected and have access limited to the study personnel.
2. Serious or severe adverse reaction to topical applications of aliquoted plasma (irritation, inflammation, infection etc.)

   1. Initial few (~3-5) topical administrations will be closely monitored in the hospital to assess for any adverse events with nursing and physician oversight.
   2. Patient/Family will be permitted to use the topical plasma independently at home only after 3-5 administrations have been monitored in hospital, parents are comfortable with storage and administration process and adverse events have been managed appropriately.
   3. In case of any adverse event such as irritation or inflammation etc. patient/family will be able to contact the responsible physician or their service at any time. Appropriate treatment strategies will be undertaken immediately for such events. Processes will be developed to prevent the adverse event from occurring in future if therapy can be continued and the event is non-fatal and non-life/limb threatening. All adverse events will be reported to the manufacturer (Canadian Blood Services).

STATISTICS

Statistical Methods Descriptive statistics for categorical and continuous variables will be used based on data points obtained and their distribution. Paired T test (or equivalent non-parametric test) will be used to determine difference in baseline and post intervention plasminogen levels at 4 weeks, 2 months, 3 months, 6 months till 24 months. A p-value of 0.05 will be considered significant. All data analyses will be conducted in Statistical software SAS version 9.4.

PLANNED PARTICIPANT ENROLLMENT One patient and 3 family members will be enrolled in this study currently. The rationale is that this is an extremely rare disorder with less than 5 patients in entire Canada and only one known patient in Saskatchewan.

DATA ACCOUNTABILITY Missing values will not be substituted by estimated values but will be treated as missing in the statistical evaluation. All data from patients randomised in the study will be included in all listings, plots, summary tables, and statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients under the age of 18 years
* Diagnosis of plasminogen deficiency (Definition: clinical presence of pseudomembranous lesions and serum plasminogen level < 50%)
* Ocular involvement (Ligneous Conjunctivitis) due to plasminogen deficiency

Exclusion Criteria:

* Patient is 18 years or older
* Patients with no plasminogen deficiency
* Patients with no ocular manifestations of plasminogen deficiency

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference in the size of pseudomembranous conjunctival lesion after 2 months of local administration of aliquoted plasma (reported as mean difference and percent difference from pre-administration size of pseudomembranous lesions ) | 24 months
  The size of pseudomembranous lesions will be measured before intervention and after 4 weeks of topical administration of aliquoted plasma in patient's conjunctiva (with/without surgical excision) 8 weeks of topical administration of plasma (with/without surgical excision). This size will be compared to the size of pseudomembranes prior to intervention. The results will be reported as mean difference and percent.
Time to change in the size of pseudomembranous lesions by 50% or greater with topical administration of aliquoted allogenic plasma in the affected conjunctiva. | 24 months. This knowledge will be aggregated in the patient data collection form
  The presence and size of pseudomembranous lesions on the patient's conjunctiva will be assessed via ophthalmologic examination every 2-7 days for first 2 months of topical application of aliquoted plasma in affected conjunctiva. The ophthalmologic assessment will then occur at increasing intervals based on the response of patient's ligneous conjunctivitis (pseudomembranous lesions) to this therapy.
  Time interval to the outcome measure (change in size of pseudomembranes) will be reported as number of days from the start of administration of aliquoted plasma.
Difference in the visual acuity of affected eye after topical administration of aliquoted allogenic plasma into affected conjunctiva. | 24 months. This information will be aggregated in data collection form
  The visual acuity in the affected eye will be assessed via ophthalmologic assessment using age-appropriate measures before intervention and on a periodic basis after the start of intervention. The difference in visual acuity before and after intervention will be reported as percent difference
Number of participants with development of strabismus or other visual defects in affected eye | 24 months. Information will be aggregated in data collection form
  Assessed via clinical ophthalmologic assessment on a periodic basis after start of administration of aliquoted plasma in patient's conjunctiva

SECONDARY OUTCOMES:
Number of participants with recurrence of pseudomembranous lesions | 24 months
Time to development of recurrence of pseudomembranous lesions in the eye undergoing intervention. | 24 months
  The time interval to development of recurrence of pseudomembranous lesions will be measured after complete resolution of pseudomembranes in affected eye.
  Time interval will be reported as number of days since complete resolution of pseudomembranes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After 12 months for 5 years
Access Criteria: Individual physicians and research groups interested in plasminogen deficiency

REFERENCES:
- [Background] Mehta R, Shapiro AD. Plasminogen deficiency. Haemophilia. 2008 Nov;14(6):1261-8. doi: 10.1111/j.1365-2516.2008.01825.x. PMID 19141167
- [Background] Schuster V, Hugle B, Tefs K. Plasminogen deficiency. J Thromb Haemost. 2007 Dec;5(12):2315-22. doi: 10.1111/j.1538-7836.2007.02776.x. Epub 2007 Sep 26. PMID 17900274
- [Background] Babcock MF, Bedford RF, Berry FA. Ligneous tracheobronchitis: an unusual cause of airway obstruction. Anesthesiology. 1987 Nov;67(5):819-21. No abstract available. PMID 3674489
- [Background] Tefs K, Gueorguieva M, Klammt J, Allen CM, Aktas D, Anlar FY, Aydogdu SD, Brown D, Ciftci E, Contarini P, Dempfle CE, Dostalek M, Eisert S, Gokbuget A, Gunhan O, Hidayat AA, Hugle B, Isikoglu M, Irkec M, Joss SK, Klebe S, Kneppo C, Kurtulus I, Mehta RP, Ornek K, Schneppenheim R, Seregard S, Sweeney E, Turtschi S, Veres G, Zeitler P, Ziegler M, Schuster V. Molecular and clinical spectrum of type I plasminogen deficiency: A series of 50 patients. Blood. 2006 Nov 1;108(9):3021-6. doi: 10.1182/blood-2006-04-017350. Epub 2006 Jul 18. PMID 16849641
- [Background] Bateman JB, Pettit TH, Isenberg SJ, Simons KB. Ligneous conjunctivitis: an autosomal recessive disorder. J Pediatr Ophthalmol Strabismus. 1986 May-Jun;23(3):137-40. doi: 10.3928/0191-3913-19860501-09. PMID 3723296
- [Background] Schuster V, Seregard S. Ligneous conjunctivitis. Surv Ophthalmol. 2003 Jul-Aug;48(4):369-88. doi: 10.1016/s0039-6257(03)00056-0. PMID 12850227
- [Background] Watts P, Agha SH, Mameesh M, Conor P, Ganesh A, Al-Mujaini A, Jewsbury H, Pathare A, Al-Rawas A. Fresh frozen plasma (Octaplas) and topical heparin in the management of ligneous conjunctivitis. J AAPOS. 2019 Feb;23(1):42-45.e1. doi: 10.1016/j.jaapos.2018.05.011. Epub 2018 Aug 27. PMID 30165199
- [Background] Ku JY, Lichtinger A, Yeung SN, Kim P, Cserti-Gazdewich C, Slomovic AR. Topical fresh frozen plasma and heparin treatment of ligneous conjunctivitis in a Canadian hospital setting. Can J Ophthalmol. 2012 Oct;47(5):e27-8. doi: 10.1016/j.jcjo.2012.03.025. Epub 2012 Jul 13. No abstract available. PMID 23036559
- [Background] Pergantou H, Likaki D, Fotopoulou M, Katsarou O, Xafaki P, Platokouki H. Management of ligneous conjunctivitis in a child with plasminogen deficiency. Eur J Pediatr. 2011 Oct;170(10):1333-6. doi: 10.1007/s00431-011-1483-9. Epub 2011 May 31. PMID 21625933
- [Background] Suzuki T, Ikewaki J, Iwata H, Ohashi Y, Ichinose A. The first two Japanese cases of severe type I congenital plasminogen deficiency with ligneous conjunctivitis: successful treatment with direct thrombin inhibitor and fresh plasma. Am J Hematol. 2009 Jun;84(6):363-5. doi: 10.1002/ajh.21402. PMID 19373890
- [Background] Shapiro AD, Menegatti M, Palla R, Boscarino M, Roberson C, Lanzi P, Bowen J, Nakar C, Janson IA, Peyvandi F. An international registry of patients with plasminogen deficiency (HISTORY). Haematologica. 2020 Mar;105(3):554-561. doi: 10.3324/haematol.2019.241158. Epub 2020 Jan 30. PMID 32001536
- [Background] Khandelwal A. Allogenic plasma aliquots for use as eye drops. Information for sponsor
- [Background] Hangul M, Tuzuner AB, Somekh I, Klein C, Patiroglu T, Unal E, Kose M. Type 1 Plasminogen Deficiency With Pulmonary Involvement: Novel Treatment and Novel Mutation. J Pediatr Hematol Oncol. 2021 May 1;43(4):e558-e560. doi: 10.1097/MPH.0000000000001951. PMID 32941296
- [Background] Rouatbi A, Chebbi A, Bouguila H. Ligneous conjunctivitis due to plasminogen deficit: Diagnostic and therapeutic approach. With literature review. J Fr Ophtalmol. 2018 Dec;41(10):916-919. doi: 10.1016/j.jfo.2018.03.012. Epub 2018 Nov 12. PMID 30442487
- [Background] Conforti FM, Di Felice G, Bernaschi P, Bartuli A, Bianco G, Simonetti A, Buzzonetti L, Valente P, Corsetti T. Novel plasminogen and hyaluronate sodium eye drop formulation for a patient with ligneous conjunctivitis. Am J Health Syst Pharm. 2016 Apr 15;73(8):556-61. doi: 10.2146/ajhp150395. PMID 27045067
- [Background] Tu Y, Gonzalez-Gronow M, Kolomeyer AM, Cohen A, Pruzon J, Milman T, Chu DS. Adult-Onset Ligneous Conjunctivitis with Detection of a Novel Plasminogen Gene Mutation and Anti-Plasminogen IgA Antibody: A Clinicopathologic Study and Review of Literature. Semin Ophthalmol. 2016;31(6):526-31. doi: 10.3109/08820538.2015.1005319. Epub 2015 Feb 12. PMID 25674820
- [Background] Ang MJ, Papageorgiou KI, Chang SH, Kohn J, Chokron Garneau H, Goldberg RA. Topical Plasminogen as Adjunctive Treatment in Recurrent Ligneous Conjunctivitis. Ophthalmic Plast Reconstr Surg. 2017 Mar/Apr;33(2):e37-e39. doi: 10.1097/IOP.0000000000000694. PMID 27065432
- [Background] Heidemann DG, Williams GA, Hartzer M, Ohanian A, Citron ME. Treatment of ligneous conjunctivitis with topical plasmin and topical plasminogen. Cornea. 2003 Nov;22(8):760-2. doi: 10.1097/00003226-200311000-00009. PMID 14576528
- [Background] Kizilocak H, Ozdemir N, Dikme G, Koc B, Atabek AA, Cokugras H, Iskeleli G, Donmez-Demir B, Christiansen NM, Ziegler M, Ozdag H, Schuster V, Celkan T. Treatment of plasminogen deficiency patients with fresh frozen plasma. Pediatr Blood Cancer. 2018 Feb;65(2). doi: 10.1002/pbc.26779. Epub 2017 Sep 6. PMID 28876531
- [Background] Park, Benjamin J., et al.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT05404932/Prot_SAP_002.pdf
  • Informed Consent Form (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT05404932/ICF_003.pdf